CLINICAL TRIAL: NCT05159713
Title: Randomized Control Trial to Evaluate the Efficacy of a Digital Mental Health Intervention Embedded in Routine Care Compared to Treatment As Usual in Adolescents and Young Adults with Moderate Depressive Symptoms
Brief Title: Study to Compare the Use of a Behavioral Health App Versus Care As Usual for 16-22 Year Olds with Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Eva Szigethy, Professor of Psychiatry and Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY21080150
Record Dates: First submitted 2021-12-01; First posted 2021-12-16 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Depression
Keywords: mobile app; digital behavioral tool; adolescent and young adult
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinician rated rated measures Children's Depression Rating Scale Revised (CDRS-R) and Clinical Global Assessment Scale (CGAS) will be completed by a blinded assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as Usual (TAU) (Other): Participants who are randomly assigned to the Treatment as Usual (TAU) group will receive standard care, which will consist of a tiered stepped care model of behavioral therapy offered by the embedded behavioral therapist at each practice as part of routine care, with the provision of augmentation of therapy (or addition of an antidepressant) at the discretion of the clinical team. Psychotropic medications at baseline and previous behavioral treatment will be recorded at baseline. Number of therapy sessions, delivery modality (face to face versus telemedicine), and addition of antidepressant or other psychotropic medication or dose change will be monitored and recorded over the study period.
  Interventions: Behavioral: Treatment as Usual
- dCBI + Treatment as Usual (Experimental): Participants randomly assigned to the intervention group (dCBI+TAU) will receive standard care and also gain access to the dCBI. The dCBI, RxWell, is a trans-Cognitive Behavioral Therapy (CBT) mobile app product addressing depression and anxiety that was developed based on standard CBT techniques.
  Interventions: Behavioral: dCBI; Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: dCBI — The dCBI, RxWell, is a trans-CBT mobile app product addressing depression and anxiety that was developed based on standard CBT techniques. RxWell provides users users with 40 brief (5-10 minute) skill building techniques for anxiety and depression. Users will have access to a goal-setting tab and "in the moment relief" section which contains over 17 techniques,14 of which are brief audios to help users engage relaxation responses. The user will be provided with the depression path, which has 40 unique techniques, and if the user expresses significant anxiety, the coach will have the ability to personalize the program by pulling in any of the 53 techniques from the anxiety path, so that the individual can utilize the proper CBT techniques that fit with their presentation.
  Arms: dCBI + Treatment as Usual
Behavioral: Treatment as Usual — Participants who are randomly assigned to the Treatment as Usual (TAU) group will receive standard care, which will consist of a tiered stepped care model of behavioral therapy offered by the embedded behavioral therapist at each practice as part of routine care, with the provision of augmentation of therapy (or addition of an antidepressant) at the discretion of the clinical team. Psychotropic medications at baseline and previous behavioral treatment will be recorded at baseline. Number of therapy sessions, delivery modality (face to face versus telemedicine), and addition of antidepressant or other psychotropic medication or dose change will be monitored and recorded over the study period.

SUMMARY:
Randomized Controlled Trial comparing a coach-enhanced digital cognitive behavioral intervention (d-CBI) (RxWell) + treatment as usual (TAU) versus TAU alone for moderate depression as determined by Patient Health Questionnaire (PHQ-9) threshold as part of routine pediatric care.

The study will be completed in pediatric practices with embedded behavioral therapists across 3 institutions (Children's Hospital of Pittsburgh, Boston Children's Hospital, Rady Children's Hospital, San Diego).

DETAILED DESCRIPTION:
After consent, participants will be further screened to determine eligibility. They will complete a brief Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM5) (SCID). If someone has been hospitalized in the past 3 months for dangerousness, or is diagnosed with severe current psychiatric disorders based on SCID V (Clinical Trials Version) for bipolar disorder, current substance misuse or dependence, or thought disorder they will not be eligible for this study and will be referred back to the clinician for further support.

PARTICIPANT PROCEDURES:

All participants who are eligible for this study, consent to participate, and are randomized to one of the two arms (dCBI+TAU or TAU) will be asked to complete self-report and blinded clinician administered measures on three occasions over 12 weeks (baseline, 6-, and 12-week time points). At enrollment and prior to randomization, each participant will be assigned a unique Study ID that will be used to code all data collected for research purposes.

Participants will be asked to complete self-report assessments via 1) self-administered completion of assessments through REDCap Cloud (i.e., online); 2) over the phone with a member of the Research Team who will enter the participant's responses into a secure web-based portal (REDCap Cloud).

ELIGIBILITY:
Inclusion Criteria:

* Age 16-22 inclusive recruited from outpatient pediatric clinic visit.
* Meeting positive screen criteria depression by PHQ-9 criteria (score greater than or equal to10).
* English-speaking (participant)
* Smart phone access

Exclusion Criteria:

* Extremely severe depression (PHQ-9 greater than 24; or active suicidal plan).
* Current dangerousness (based on Treatment for Adolescents for Depression Study (TADS) study criteria, 2004). Hospitalized for dangerousness within 3 months; Suicide attempt requiring medical attention within 3 months.
* Severe, current psychiatric disorders based on SCID V (Clinical Trials Version) for bipolar disorder, current substance misuse or dependence, thought disorder. Research coordinators who are trained to fidelity threshold will complete this measure with the patient.

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 185 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Change in depression severity | 12 weeks
  Children's Depression Rating Scale-Revised (CDRS-R) will be administered by a blinded rater from baseline up to 12 weeks after baseline to evaluate the change in depression severity.
  The CDRS-R is a 17-item interview, which score can add up to between 17 and 113. A score of greater than or equal to 40 indicates depressive symptomatology, and a score of less than or equal to indicates remission.

SECONDARY OUTCOMES:
Change in depression severity; evidence of passive suicidal ideation | 12 weeks
  Patient Health Questionnaire (PHQ-9) will be utilized to measure change in depression severity and evidence of passive suicidal ideation from baseline up to 12 weeks after baseline.
  The PHQ-9 is a 9 item questionnaire. Scores can range from 0-27. A score of 0-4 indicates no depressive symptoms; 5-9 indicates mild depressive symptoms; 10-19 indicates moderate depressive symptoms; 20-27 indicates severe depressive symptoms.
Change in anxiety severity | 12 weeks
  Generalized Anxiety Disorder (GAD7) will be utilized to measure change in anxiety severity from baseline up to 12 weeks after baseline.
  GAD-7 is a 7 item questionnaire. Scores range from 7-21. Total scores of 0-4 indicates no anxiety; 5-9 mild anxiety; 10-14 moderate anxiety; greater than or equal to 15 indicates severe anxiety.
Change in quality of life | 12 weeks
  Satisfaction with Life Scale (SWLS) will be utilized to measure change in quality of life from baseline up to 12 weeks after baseline.
  SWLS is a five item measure with a maximum score of 35. Higher score correlate with higher satisfaction of life. Scores 31-35 extremely satisfied. Scores less than 9 indicate extremely dissatisfied.
Change in general level of functioning | 12 weeks
  Children's Global Assessment Scale (CGAS) blinded clinician rater will be utilized to measure the level of general functioning from baseline up to 12 weeks after baseline.
  CGAS scores range from 1-100 with 100-91 associated with superior functioning and 31-40 with major impairment in functioning in several areas, and unable to function in one of those areas.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Szigethy, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - Rady Children's Hospital - San Diego, San Diego, California
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared. Data is shared at the aggregate level.

REFERENCES:
- [Derived] Szigethy E, Wolfson D, Sinclair-McBride K, Williams K, Jhe G, Lee EH, Bialostozky M, Wallace M, Bhatnagar S, Demaso DR, Yealy DM, Hollenbach K. Efficacy of a digital mental health intervention embedded in routine care compared with treatment as usual in adolescents and young adults with moderate depressive symptoms: protocol for randomised controlled trial. BMJ Open. 2023 Mar 31;13(3):e067141. doi: 10.1136/bmjopen-2022-067141. PMID 37001917